CLINICAL TRIAL: NCT05129332
Title: The Impact of Vaginal Dilator Therapy on Pain Scores and Sexual Function Among Women With Gynecologic and Breast Cancers Experiencing Dyspareunia: a Randomized Controlled Trial
Brief Title: Vaginal Dilator Therapy Among Women With Gynecologic and Breast Cancers Experiencing Dyspareunia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study was stopped as Fellow was unable to committ to enrollment and study due to time constraints
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Jason D. Wright, Sol Goldman Associate Professor of Gynecologic Oncology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAT8915
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Dyspareunia
Keywords: Painful Intercourse; Sexual Dysfunction; Vaginal Dilator; Vaginal Moisturizer
MeSH Terms: conditions — Dyspareunia; Sexual Dysfunction, Physiological | interventions — Vitamin E; Coconut Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Vaginal Dilator Intervention (Experimental): Patients assigned to the vaginal dilator group will be provided the device, vaginal moisturizer, an adherence calendar, and standardized verbal and written instructions from a trained health professional to apply the moisturizer and use the dilator for 15 minutes daily. Standard medical grade vaginal dilators and pure Vitamin E oil will be provided for each study participant. They have the option of purchasing a dilator and/or moisturizer of a similar nature if they choose to.
  Interventions: Other: Vaginal Moisturizer; Device: Vaginal Dilator
- Control (Vaginal Moisturizer Only) (Other): Patients assigned to vaginal moisturizer alone will receive pure Vitamin E oil and similar standardized instructions on daily use and an adherence calendar. They will apply a dime-sized amount of Vitamin E oil every day. They have the option of purchasing their own moisturizer if they choose to.
  Interventions: Other: Vaginal Moisturizer

INTERVENTIONS:
Other: Vaginal Moisturizer — Natural oil-based vaginal moisturizers, like Vitamin E Oil or Coconut Oil, will be applied topically (dime-size amount) on the labia externally and vagina internally nightly, but at least 3 times per week.
  Other Names: Vitamin E Oil; Coconut Oil
Device: Vaginal Dilator — Vaginal dilator will be inserted vaginally and used daily, but at least 3 times per week.
  Arms: Vaginal Dilator Intervention

SUMMARY:
In this randomized controlled trial, the investigators will assess the difference in mean patient-reported pain scores and sexual function between women with gynecologic or breast cancers experiencing dyspareunia (painful intercourse) who are assigned to vaginal dilator use with vaginal moisturizer (Intervention Group, n = 29) compared to vaginal moisturizer alone (Control Group, n = 29) over 16 weeks.

DETAILED DESCRIPTION:
Between 2012 and 2016, approximately 94,000 women were diagnosed with a gynecologic cancer annually and over 1.2 million women with breast cancer between 2013 and 2017. It is well known that gynecologic and breast cancers, and their treatments including surgery, adjuvant chemotherapy and endocrine therapy, and radiation, result in significant effects on the female reproductive system which can lead to sexual dysfunction. In the U.S., sexual dysfunction among gynecologic oncology patients has been reported to be as high as 90%, and over 70% among breast cancer patients. Patients who receive chemotherapy and/or endocrine therapy commonly experience dyspareunia, vaginal dryness, and challenges with desire and orgasm due to a low estrogen state. In fact, among patients with breast cancer, unaddressed sexual side effects from adjuvant endocrine therapy are one reason for early discontinuation. Hysterectomy and oophorectomy, including for ovarian cancer risk-reduction, can cause similar physical symptoms in addition to psychologic effects like anxiety related to sexual intercourse.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* English or Spanish speaking
* Patients currently or previously treated for:

  * Gynecologic cancer (surgery, chemotherapy, adjuvant vaginal brachytherapy)
  * Breast cancer (chemotherapy, aromatase inhibitors, or selective estrogen receptor modulators; surgical menopause)
* Current desire for penetrative sexual activity
* Endorsement of at least one of the following in the last 6 months:

  * Dyspareunia during penetrative sexual activity
  * Reported sensation of penetrative object (partner's penis, sex toy) not fitting in the vagina
  * Avoidance of penetrative sexual activity due to fear of pain
* Physically able to insert a vaginal dilator by themselves
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with prior primary or upfront pelvic radiation
* Patients with whole pelvic radiation at any time
* Patients with a history of chronic pelvic pain
* Patients with vulvodynia as noted on baseline pelvic exam with > 5/10 pain score during an external exam with a cotton swab
* Patients with prior vaginal dilator use for any indication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Difference in Mean Patient-Reported Pain Scores During Sexual Activity | Up to 16 weeks
  The difference in mean patient-reported pain scores will be calculated, during penetrative sexual activity before and after randomization to vaginal dilator use with vaginal moisturizer or vaginal moisturizer alone. Pain scores will be assessed using a 10cm vial analog scale (VAS), in which 0 indicates no pain and 10 indicates most pain (worst outcome).

SECONDARY OUTCOMES:
Difference in Mean Patient-Reported Pain Scores During Speculum Exam | Up to 16 weeks
  The difference in mean patient-reported pain scores will be calculated, during speculum exam before and after randomization to vaginal dilator use with vaginal moisturizer or vaginal moisturizer alone. Pain scores will be assessed using a 10cm vial analog scale (VAS), in which 0 indicates no pain and 10 indicates most pain (worst outcome).

OTHER OUTCOMES:
Sexual Function based on the PROMIS SexFS Score (Version 2.0) | Up to 16 weeks
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Sexual Function (SexFS) assesses over the last 30 days interest in sexual activity, lubrication, vaginal discomfort, clitoral discomfort, labial discomfort, erectile function, orgasm ability, orgasm pleasure and is customizable so that study designers can select relevant domains and items for their study. Raw scores can range from 2 to 10 ("very" or "very much"), which is then converted to a T-score found in the appendix of the survey. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore a person with a T-score of 40 is one SD below the mean. The standardized T-score is reported as the final score for each participant for each domain.

CONTACTS AND LOCATIONS:
Overall Officials: Jason D. Wright, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Irving Medical Center / NewYork-Presbyterian Hospital, New York, New York
  - Women & Infants Hospital of Rhode Island / Brown University, Providence, Rhode Island